CLINICAL TRIAL: NCT00581347
Title: Primary Care and Adolescent Immunization for Rochester
Acronym: PCAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PCAIR; OPP-P-2006-24
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Adolescent Immunizations; Preventive Care

ARMS (2):
- Outreach (Other): Receives outreach services
  Interventions: Other: outreach services
- Standard of Care (No Intervention): Receives standard medical care provided by primary care practice.

INTERVENTIONS:
Other: outreach services — Tracking/reminder/recall/home visit strategy.
  Arms: Outreach

SUMMARY:
This study will examine whether the implementation of an outreach program that employs a tracking/reminder/recall/home visiting strategy will have any impact on receipt of immunizations and preventive care among urban adolescents.

DETAILED DESCRIPTION:
Outreach workers will be placed at 9 primary care pediatric and family medicine practices throughout one urban area. Adolescent patients at these 9 practices will be identified and then randomized into two groups; (1) those receiving outreach intervention during Year 1 of the study and (2) those receiving outreach intervention during Year 2 of the study. Randomization will be stratified by practice site, patient age, and patient gender.

After randomization, the list of Year 1 subjects will be distributed to the appropriate outreach worker. The outreach worker will track the immunization status of 11-15yo patients within their practice, identify patients who are eligible for but have not yet received immunizations recommended for their age group (MMR, Varicella, Hepatitis B, HPV, Meningococcal Conjugate, Tdap) and/or a well child visit within the past year, and then attempt to connect these patients with medical care through three levels of outreach activity. First level of outreach activity involves contacting the parent/guardian of the patient by telephone. Outreach workers will attempt to inform patient's parent/guardian of needed immunizations/preventive visit and facilitate the scheduling of a medical appointment. If unable to successfully complete the task through telephone contact, outreach workers will initiate the second level of outreach activity - contact by mail. If contact by mail is unsuccessful, the third and most intense level of outreach activity will be implemented. The outreach worker will attempt to notify the patient's parent/guardian of need for immunization/preventive appointment by visiting the patient's listed home address. During this visit, the outreach worker will attempt to inform the parent/guardian of recommended immunizations, provide information pertaining to these immunizations, facilitate appointment scheduling, and assist patient in compliance with scheduled medical appointment

Interventions directed towards the subjects of the Year 1 group will cease after 15 months of outreach activity. A chart review of intervention and control groups will be conducted to determine immunization and well child visit rates within the two groups. At this time, the tracking/reminder/recall/home visiting strategy employed with the Year 1 group will be repeated for Year 2 subjects.

ELIGIBILITY:
Inclusion Criteria:

* 11-15 years of age
* receive medical care at one of the 9 pediatric or family medicine practices identified as study sites

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7546 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Szilagyi PG, Humiston SG, Gallivan S, Albertin C, Sandler M, Blumkin A. Effectiveness of a citywide patient immunization navigator program on improving adolescent immunizations and preventive care visit rates. Arch Pediatr Adolesc Med. 2011 Jun;165(6):547-53. doi: 10.1001/archpediatrics.2011.73. PMID 21646588

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target population was teens with birthdates between 7/1/92 & 6/30/97 at 8 practices in Rochester, NY. 2 methods were used to identify eligible adolescents;(1)2 insurance plans in the region provided a list of all their pts at these practices. (2)2 practices added to the list all teens who made a visit within 2 years of the study start date.
Pre-assignment Details: We preformed a stratified random sample, allocating all adolescents to either an intervention or standard of care group (using SAS 9.1). We stratified by practice, age and gender. For families with 2 or more eligible siblings, we assigned all siblings to the same group. Healthcare providers were unaware of group assignment.
Groups:
- Outreach: The intervention consisted of a tiered protocol, with each step being more intensive and targeting a progressively smaller proportion of adolescents who remained behind in immunizations. The intervention was delivered by trained patient immunization navigators.
  Step 1- Patient tracking: We used a web-based database to track the adolescents in the intervention group, record immunizations and preventive visits, and document tasks they performed.
  Step 2: Reminders and recall: The navigators performed reminder/recall for adolescents who were eligible for either a vaccination or a preventive care visit. They attempted to contact families by telephone and mail.
  Step 3: Home visits: If adolescents remained unvaccinated despite the above steps, the navigators performed a home visit to further assess barriers, promote the importance of preventive care, and encourage families to make appointments.
- Standard of Care: Control subjects received standard of care. All practices routinely sent letter or telephone reminders to families who had upcoming scheduled visits, but none used active reminder/recall based on vaccinations.
Period: Overall Study
Arm/Group | Outreach | Standard of Care
Started | 3839 | 3707
Completed | 3839 | 3707
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Outreach | Standard of Care | Total
Number analyzed (Participants) | 3839 | 3707 | 7546
Age, Customized [Number; unit: participants]
  11 years old | 784 | 757 | 1541
  12 years old | 743 | 701 | 1444
  13 years old | 714 | 686 | 1400
  14 years old | 781 | 758 | 1539
  15 years old | 817 | 805 | 1622
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1903 | 1849 | 3752
  Male | 1936 | 1858 | 3794

OUTCOME MEASURES:

1. Primary Outcome: Receipt of Adolescent Immunization at End of Study Period (Tdap, Menactra, HPV)
Description: We compared the number of participants in the intervention group who received vaccinations for Tdap, Menactra, and (for girls only) HPV at the end of the study period versus those in the control group.
Time Frame: 15 months
Measure: Number; unit: participants
Arm/Group | Outreach | Standard of Care
Number analyzed (Participants) | 3839 | 3707
participants
  Tdap | 1091 | 885
  Menactra | 1783 | 1367
  HPV 1 | 634 | 453
  HPV 2 | 827 | 560
  HPV 3 | 671 | 432

2. Secondary Outcome: Receipt of a Well Child Visit Within a 12 Month Period
Description: We compared the number of participants in the intervention group who received a well child visit within a 12 month period versus those in the control group.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Outreach | Standard of Care
Number analyzed (Participants) | 3839 | 3707
participants | 2609 | 2045

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Outreach | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/3839 | 0/3707
Other Adverse Events (participants affected / at risk) | 0/3839 | 0/3707
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Outreach (N=3839) | Standard of Care (N=3707)
HIPAA violation (Social circumstances) | 0 (0) | 0/0 (0) — An unauthorized disclosure of personally-identifiable health information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No